CLINICAL TRIAL: NCT06498089
Title: A Randomized, Controlled, Open-label, Multicenter Clinical Trial Comparing the Efficacy and Safety of a Precision Treatment Regimen Based on Clinical-molecular Phenotypes with a Conventional Treatment Regimen in the Treatment of Patients with Active Takayasu's Arteritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2024-200R
Record Dates: First submitted 2024-06-29; First posted 2024-07-12 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Takayasu Arteritis
Keywords: Precise treatment; Clinical-molecular phenotype
MeSH Terms: conditions — Takayasu Arteritis | interventions — Prednisone; Glucocorticoids; Methotrexate; tocilizumab; tofacitinib; Adalimumab

STUDY DESIGN:
Intervention Model Description: This study was a randomized, controlled study, including two arms.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The precise therapy arm (Experimental): Patients will be given treatment based on their clinical-molecular phenotype according to a predesigned scheme:
  1. Patients in constitutional type will be given treatments with GCs combined with TCZ and MTX.
  2. Patients in vascular inflammation type without IL-6 and TNF-α elevation will be given treatments with GCs combined with TOF.
  3. Patients in vascular inflammation type with IL-6 elevation will be given treatments with GCs combined with TCZ and MTX.
  4. Patients in vascular inflammation type with TNF-α elevation will be given treatments with GCs combined with ADA and MTX.
  Interventions: Drug: Prednisone; Drug: Methotrexate; Drug: Tocilizumab; Drug: Tofacitinib; Drug: Adalimumab
- The traditional therapy arm (Active Comparator): Patients will be given traditional treatment based on their clinical-molecular phenotype according to a predesigned scheme.
  Interventions: Drug: Prednisone; Drug: Methotrexate

INTERVENTIONS:
Drug: Prednisone — This drug will be used in both arms. Patients' initial daily prednisone dose will be calculated according to their weights (0.6mg * weight(kg), maximum 50mg/day), and then tapered gradually during the study course.
  Other Names: Glucocorticoids
Drug: Methotrexate — This drug will be used in the traditional arm. A dose of 15mg per week will be used.
  Other Names: MTX
Drug: Tocilizumab — This drug will be used in the precise treatment arm. For patients in constitutional type a dose (8mg/kg weight) will be used every 2 weeks (iv drip) for 12 weeks, then a dose (8mg/kg weight) will be used every 4 weeks (iv drip). For patients in vascular inflammation type, a dose (8mg/kg weight) will be used every 4 weeks (iv drip).
  Other Names: TCZ
  Arms: The precise therapy arm
Drug: Tofacitinib — This drug will be used in the precise treatment arm. A sustained release tablet will be used (11mg per day).
  Other Names: TOF
  Arms: The precise therapy arm
Drug: Adalimumab — This drug will be used in the precise treatment arm. A dose of 40mg (ih) will used every 2 weeks.
  Other Names: ADA
  Arms: The precise therapy arm

SUMMARY:
This study aimed to compare the efficacy and safety of a precision treatment regimen based on clinical-molecular phenotypes with a conventional treatment regimen in the treatment of patients with active Takayasu's arteritis based on a randomized, controlled, open-label, multicenter study.

DETAILED DESCRIPTION:
1. This study is a randomised, controlled, open-label, evaluator-blinded, multicentre clinical trial with a 14-month (56-week) study period: a 6-month (0-24 weeks) induction remission period and an 8-month (24-56 weeks) maintenance remission period;
2. Subjects with aortitis who meet the entry criteria will be randomised and divided 1:1 into the precision therapy group and the conventional therapy group. The precision therapy group will be stratified according to the clinical-molecular phenotypes, and at the end of 6 months, if subjects achieve clinical remission and the amount of GCs is reduced to 7.5 mg/day for 4 weeks, they will enter into the maintenance period and continue with the original regimen; if they do not meet this, they will be withdrawn from the study;
3. The study adopts a superiority design, the primary study objective is to assess the efficacy of the two groups at the end of six months, and the secondary study objectives are to assess the efficiency of the two groups at the end of 12 months, relapse rate, safety, cumulative hormone dose, vascular imaging changes, changes in cytokine profiles, etc.
4. According to their new-onset symptoms at baseline or within past three months, the patients were divided into two clinical phenotypes: ①constitutional type: patients with constitutional symptoms, such as fever, fatigue, weakness, and weight loss, without any symptoms of organ ischemia, and at least 4 of the following indicators were above normal upper limits: ESR, CRP, C3, PLT, IL-6, C4, IgG; ②vascular inflammation type: patients with vascular-associated symptoms, such as carotidynia, angina, dizziness, and limb claudication, regardless of the constitutional symptoms or ischemic symptoms.

ELIGIBILITY:
Inclusion Criteria:

1) Meet the 2022 ACR/EULAR classification criteria for aortitis; 2) Women or men aged 18-65 years; 4) Be in active disease: a National Institutes of Health (NIH) score of ≥2; 5) Females with negative serum or urine pregnancy test results and no plans to have children during the clinical trial; (6) If the patient is taking prednisone or its equivalent, the pre-enrolment dose does not exceed 0.6 mg/kg/day and the dose has been stable for at least 4 weeks; 7) If the patient is receiving other medications for aortitis that are inconsistent with the assigned regimen, discontinuation is required for ≥4 weeks for methotrexate, azathioprine, mycophenolate mofetil, cyclosporine, and tacrolimus; for leflunomide, discontinuation is required for 11 days if elimination methods are used (kolexanil or activated charcoal), or ≥8 weeks if elimination is not used; for cyclophosphamide, discontinuation is required for ≥6 months; for biologics, stopping for ≥ 3 weeks is required for etanercept, ≥ 4 weeks for IL-6 receptor antagonists and tumour necrosis factor inhibitors, and ≥ 6 months for rituximab.

8)For patients with no obvious active tuberculosis lesions but elevated T-spot, it is recommended that infectious specialists evaluate them, and preventive anti-tuberculosis therapy should be performed first if necessary. After T-spot declines, researchers will assess the relevant risks before deciding whether they are suitable to participate in this study, and continue preventive anti-tuberculosis therapy for a total of 9 months.

9)For patients with HBV, if the viral replication was detected, it is recommended to take anti-viral treatment for 2-4 weeks, and researchers will evaluate whether they are suitable to participate in this study when no DNA replication is detected.

Exclusion Criteria:

1. Presence of organ failure;
2. undergoing haemodialysis or major surgery (grade III and above) within 3 months;
3. the presence of other autoimmune diseases;
4. severe, progressive organ damage;
5. Subjects with other comorbidities that may result in the need for additional moderate to high doses of glucocorticoids (prednisone ≥ 10 mg/day or equivalent doses of prednisone equivalents) during the study period;
6. Have a history of malignancy;
7. Have any serious acute or chronic infection, including hepatitis B surface antigen positive, active tuberculosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness rate | 6 months
  Effectiveness is defined if patients meet the following three in criteria ①-④ and criteria ⑤.
  * No systemic symptoms such as fever, malaise, or wasting;
    * No new onset of vascular symptoms and signs;
      * Normal blood sedimentation (in case of abnormality, it is necessary to exclude non-disease active factors and to review and evaluate with the review value); ④ Imaging: no progression of primary vascular lesions or new vascular lesions; ⑤ Glucocorticoids are reduced to 7.5mg/day and maintained for at least 4 weeks.

SECONDARY OUTCOMES:
Effectiveness rate | 12 months
  * No systemic symptoms such as fever, malaise, or wasting;
    * No new onset of vascular symptoms and signs;
      * Normal blood sedimentation (in case of abnormality, it is necessary to exclude non-disease active factors and to review and evaluate with the review value); ④ Imaging: no progression of primary vascular lesions or new vascular lesions; ⑤ Glucocorticoids are reduced to 5mg/day and maintained for at least 4 weeks.
Relapse rate | 12 months
  The relapse is defined as disease re-activation after remission. Disease activity is assessed according to NIH criteria. NIH≥2 is considered active status.
  NIH criteria includes:
  * Systemic symptoms, such as fever, skeletal and muscular symptoms;
    * Blood sedimentation (erythrocyte sedimentation rate, ESR) >20mm/H; ③ Characteristics of vascular ischaemia or inflammation: e.g. intermittent claudication, diminished or absent pulse, vascular murmur, vascular pain blood pressure asymmetry; ④Abnormalities of angiography.
Time to the first relapse | 12 months
  The first time to develop relapse during 12 months' treatment.
Adverse events | 12 months
  The occurrence of adverse events and the corresponding rate.
Vascular imaging changes | 12 months
  New vascular lesions, vascular thickness changes, vascular stenosis changes and vascular dilation changes upon MRA or CTA.
Cytokine changes | 12 months
  Changes of different cytokine profiles, including interleukin levels, chemotactic protein levels, fibrotic marker levels. The spepcific parameters include PTX3, IL6, IFN-g,TNFa, IL8, IL10, IL17, YKL40, CCL22, IL16, CCL2, CCL5, VEGF-A, PDGF-AB, FGF2, MMP1,MMP2, MMP3, MMP9,Leptin, PCSK5, FABP3, GPNMB.
Improvement of Visual Analog Score for pain | 12 months
  Visual Analog Score for pain score ranges from 0 to 10, higher scores indicate a worse outcome.
Improvement of 36-Item Short Form Survey | 12 months
  The 36-Item Short Form Survey score ranges from 0 to 800, higher scores indicate a better outcome.
Improvement of Functional Assessment of Chronic Illness Therapy - Fatigue | 12 months
  The Functional Assessment of Chronic Illness Therapy - Fatigue score ranges from 0 to 52, higher socres indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, PhD, Study Chair — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
No appliable